CLINICAL TRIAL: NCT03269110
Title: Folic Acid Clinical Trial: Follow up of Children (FACT 4 Child)
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CTO 816
Record Dates: First submitted 2017-08-10; First posted 2017-08-31 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder; Asthma; Executive Dysfunction; Emotional Problem; Behavioural Problem; Pre-Eclampsia; Death
Keywords: neurological; autism; ASD; behaviour; folic acid; pre-eclampsia; asthma; executive function
MeSH Terms: conditions — Autism Spectrum Disorder; Asthma; Mental Disorders; Pre-Eclampsia; Death; Neurologic Manifestations; Autistic Disorder; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother and child(ren): FACT 4 Child is the post-delivery follow-up of the offspring born to FACT mothers once these children are between the age of 4 - 6 years.
  Interventions: Diagnostic Test: SRS 2, CBCL, BRIEF-P

INTERVENTIONS:
Diagnostic Test: SRS 2, CBCL, BRIEF-P — This study does not involve an intervention.

SUMMARY:
FACT 4 Child is a follow up study of mothers who participated in the Folic Acid Clinical Trial (NCT01355159) and their children at 4-6 years of age to determine the effect of high dose folic acid supplementation on social impairments associated with Autism Spectrum Disorders (ASDs), and deficiencies in a range of executive function and emotional and behavioural problems in young children, and the risk of death.

DETAILED DESCRIPTION:
The Folic Acid Clinical Trial (FACT) was developed to conclusively determine the effect of high dose folic acid supplementation in pregnancy on the prevention of preeclampsia in a randomized controlled trial (RCT) design.

The primary objective of the FACT 4 Child study is to examine the effect of maternal folic acid supplementation in pregnancy on the risk of social impairments, as well as executive function, emotional and behavioural problems associated with Autism Spectrum Disorders (ASD) and other developmental disorders, and death in offspring aged 4-6 y of mothers recruited to the CIHR funded FACT.

The effect of folic acid supplementation throughout pregnancy may potentially have an impact on both the mother and her offspring, which highlights the importance and relevance of this study to the management of women with preeclampsia. Results of this study will allow care providers to have the evidence of potential effects of high dose folic acid that can then be discussed; allowing women to make an informed choice about their management and care.

ELIGIBILITY:
Inclusion Criteria:

1. Capability of participant to comprehend and comply with study requirements
2. Mother participated in FACT

Exclusion Criteria:

1. Confirmed spontaneous termination (miscarriage) or elective termination or stillborn
2. Confirmed death of offspring at 6 weeks postpartum and/or at discharge from hospital

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: FACT 4 Child is the post-delivery follow-up of offspring born to FACT mothers once children reach the age of 4 years. Women in FACT and their children, will be invited to participate in FACT 4 Child.
Sampling Method: Non-Probability Sample
Enrollment: 664 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Neurocognitive disability | From six weeks of age to date of data collection taken at one time point between the ages of 4 to 6 years.
  The primary outcome is a competing composite endpoint of neurocognitive disability and death. Neurocognitive disability is a composite outcome related to social impairments, executive function, emotional and behavioural problems which have been associated with Autism Spectrum Disorder (ASD). It will be defined by an abnormal score on any of three standardized and validated assessment tools: SRS-2 BRIEF-P, or CBCL which will be administered to the parents of children aged 4-6 years. Deaths reported between 6 weeks to 4-6 years of age will be recorded as a competing event and treated as part of the primary endpoint.

SECONDARY OUTCOMES:
Severe Morbidity | From six weeks of age to date of data collection taken at one time point between the ages of 4 to 6 years.
  Secondary outcomes to be assessed in FACT 4 Child include severe morbidity of FACT offspring, captured by the Mother-Child Health Survey at the age of 4 - 6 years, including incidence of: Severe morbidity defined by any illnesses during the previous years that has necessitated hospitalization or medication/treatment for >2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Walker, MD, Principal Investigator — The Ottawa Hospital
Locations (58):
- Australia (6):
  - Nepean, Penrith, New South Wales
  - Townsville, Douglas, Queensland
  - Ipswich, Ipswich, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - Royal Women's, Parkville, Victoria
  - Sunshine, St Albans, Victoria
- Canada (18):
  - Calgary Foothills Medical Center, Calgary, Alberta
  - Edmonton Lois Hole Hospital for Women, Edmonton, Alberta
  - St-Paul's Hospital, Vancouver, British Columbia
  - Winnipeg University of Manitoba, Winnipeg, Manitoba
  - Fredericton Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - Moncton Hospital, Moncton, New Brunswick
  - St-John's Women's Health Centre, St. John's, Newfoundland and Labrador
  - Hamilton McMaster University, Hamilton, Ontario
  - Kingston, Kingston, Ontario
  - London, London, Ontario
  - The Ottawa Hospital, General Campus, Ottawa, Ontario
  - The Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences, Toronto, Ontario
  - Quebec City (CHUL) Centre Hospitalier Universitaire, Montreal, Quebec
  - Sainte-Justine, Montreal, Quebec
  - St-Mary's Hospital, Montreal, Quebec
  - St-Luc, Montreal, Quebec
  - Regina Qu'Appelle Health Region, Regina, Saskatchewan
- Jamaica (3):
  - Jubilee, Kingston
  - Spanishtown, Kingston
  - University of West Indies, Kingston
- United Kingdom (31):
  - Hinchingbrooke, Huntingdon, Cambridgeshire
  - Leighton, Crewe, Cheshire
  - Darlington Memorial Hospital, Darlington, County Durham
  - Fairfield, Bury, Lancashire
  - Rochdale, Rochdale, Lancashire
  - Lincolnshire, Lincoln, Lincolnshire
  - West Middlesex University Hospital, Isleworth, Middlesex
  - Wansbeck General Hospital, Ashington, Northumberland
  - St George's Hospital, London, Tooting
  - Gateshead Queen Elizabeth Hospital, Gateshead, Tyne and Wear
  - South Tyneside Distrcit Hospital, South Shields, Tyne and Wear
  - Blackburn, Blackburn
  - Burnley, Burnley
  - Cumberland Infirmary Carlisle, Carlisle
  - North Manchester, Crumpsall
  - North Durham, Durham
  - Guy's and St. Thomas, London
  - South Tees Hospital, Middlesbrough
  - Newcastle upon Tyne Hospitals, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Norfolk & Norwich, Norwich
  - Nottingham City Hospital, Nottingham
  - Nottingham Queens Medical Centre, Nottingham
  - Oldham, Oldham
  - North Tees Hospital, Stockton
  - Sunderland Royal Hospital, Sunderland
  - Hillingdon Hospital, Uxbridge
  - Warrington Hospital, Warrington
  - West Cumberland Hospital, Whitehaven
  - 49 Marine Avenue, Whitley Bay
  - Royal Wolverhampton - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christensen DL, Baio J, Van Naarden Braun K, Bilder D, Charles J, Constantino JN, Daniels J, Durkin MS, Fitzgerald RT, Kurzius-Spencer M, Lee LC, Pettygrove S, Robinson C, Schulz E, Wells C, Wingate MS, Zahorodny W, Yeargin-Allsopp M; Centers for Disease Control and Prevention (CDC). Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years--Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2012. MMWR Surveill Summ. 2016 Apr 1;65(3):1-23. doi: 10.15585/mmwr.ss6503a1. PMID 27031587
- [Background] Knapp M, Romeo R, Beecham J. Economic cost of autism in the UK. Autism. 2009 May;13(3):317-36. doi: 10.1177/1362361309104246. PMID 19369391
- [Background] Buescher AV, Cidav Z, Knapp M, Mandell DS. Costs of autism spectrum disorders in the United Kingdom and the United States. JAMA Pediatr. 2014 Aug;168(8):721-8. doi: 10.1001/jamapediatrics.2014.210. PMID 24911948
- [Background] McQuiston S, Kloczko N. Speech and language development: monitoring process and problems. Pediatr Rev. 2011 Jun;32(6):230-8; quiz 239. doi: 10.1542/pir.32-6-230. No abstract available. PMID 21632874
- [Background] Waddell C, McEwan K, Shepherd CA, Offord DR, Hua JM. A public health strategy to improve the mental health of Canadian children. Can J Psychiatry. 2005 Mar;50(4):226-33. doi: 10.1177/070674370505000406. PMID 15898462
- [Background] Repchinsky C. CPS 2008: Compendium of Pharmaceuticals and Specialties : The Canadian Drug Reference for Health Professionals. United States: Canadian Pharmacists Association, 2008.
- [Background] ACOG Committee on Practice Bulletins--Obstetrics. ACOG practice bulletin. Diagnosis and management of preeclampsia and eclampsia. Number 33, January 2002. Obstet Gynecol. 2002 Jan;99(1):159-67. doi: 10.1016/s0029-7844(01)01747-1. PMID 16175681
- [Background] Oakley GP Jr. Elimination of folic acid-preventable neural tube defects. Am J Prev Med. 2008 Dec;35(6):606-7. doi: 10.1016/j.amepre.2008.09.017. No abstract available. PMID 19000851
- [Background] Wilson RD; GENETICS COMMITTEE; MOTHERISK. RETIRED: Pre-conceptional vitamin/folic acid supplementation 2007: the use of folic acid in combination with a multivitamin supplement for the prevention of neural tube defects and other congenital anomalies. J Obstet Gynaecol Can. 2007 Dec;29(12):1003-1013. doi: 10.1016/S1701-2163(16)32685-8. English, French. PMID 18053387
- [Background] Suren P, Roth C, Bresnahan M, Haugen M, Hornig M, Hirtz D, Lie KK, Lipkin WI, Magnus P, Reichborn-Kjennerud T, Schjolberg S, Davey Smith G, Oyen AS, Susser E, Stoltenberg C. Association between maternal use of folic acid supplements and risk of autism spectrum disorders in children. JAMA. 2013 Feb 13;309(6):570-7. doi: 10.1001/jama.2012.155925. PMID 23403681
- [Background] Schmidt RJ, Tancredi DJ, Ozonoff S, Hansen RL, Hartiala J, Allayee H, Schmidt LC, Tassone F, Hertz-Picciotto I. Maternal periconceptional folic acid intake and risk of autism spectrum disorders and developmental delay in the CHARGE (CHildhood Autism Risks from Genetics and Environment) case-control study. Am J Clin Nutr. 2012 Jul;96(1):80-9. doi: 10.3945/ajcn.110.004416. Epub 2012 May 30. PMID 22648721
- [Background] Schmidt RJ, Hansen RL, Hartiala J, Allayee H, Schmidt LC, Tancredi DJ, Tassone F, Hertz-Picciotto I. Prenatal vitamins, one-carbon metabolism gene variants, and risk for autism. Epidemiology. 2011 Jul;22(4):476-85. doi: 10.1097/EDE.0b013e31821d0e30. PMID 21610500
- [Background] Villamor E, Rifas-Shiman SL, Gillman MW, Oken E. Maternal intake of methyl-donor nutrients and child cognition at 3 years of age. Paediatr Perinat Epidemiol. 2012 Jul;26(4):328-35. doi: 10.1111/j.1365-3016.2012.01264.x. Epub 2012 Mar 14. PMID 22686384
- [Background] Forns J, Torrent M, Garcia-Esteban R, Caceres A, Pilar Gomila M, Martinez D, Morales E, Julvez J, Grimalt JO, Sunyer J. Longitudinal association between early life socio-environmental factors and attention function at the age 11 years. Environ Res. 2012 Aug;117:54-9. doi: 10.1016/j.envres.2012.04.007. Epub 2012 May 18. PMID 22608140
- [Background] Chatzi L, Papadopoulou E, Koutra K, Roumeliotaki T, Georgiou V, Stratakis N, Lebentakou V, Karachaliou M, Vassilaki M, Kogevinas M. Effect of high doses of folic acid supplementation in early pregnancy on child neurodevelopment at 18 months of age: the mother-child cohort 'Rhea' study in Crete, Greece. Public Health Nutr. 2012 Sep;15(9):1728-36. doi: 10.1017/S1368980012000067. Epub 2012 Feb 8. PMID 22314109
- [Background] Roth C, Magnus P, Schjolberg S, Stoltenberg C, Suren P, McKeague IW, Davey Smith G, Reichborn-Kjennerud T, Susser E. Folic acid supplements in pregnancy and severe language delay in children. JAMA. 2011 Oct 12;306(14):1566-73. doi: 10.1001/jama.2011.1433. PMID 21990300
- [Background] Steenweg-de Graaff J, Roza SJ, Steegers EA, Hofman A, Verhulst FC, Jaddoe VW, Tiemeier H. Maternal folate status in early pregnancy and child emotional and behavioral problems: the Generation R Study. Am J Clin Nutr. 2012 Jun;95(6):1413-21. doi: 10.3945/ajcn.111.030791. Epub 2012 May 9. PMID 22572645
- [Background] Roza SJ, van Batenburg-Eddes T, Steegers EA, Jaddoe VW, Mackenbach JP, Hofman A, Verhulst FC, Tiemeier H. Maternal folic acid supplement use in early pregnancy and child behavioural problems: The Generation R Study. Br J Nutr. 2010 Feb;103(3):445-52. doi: 10.1017/S0007114509991954. Epub 2009 Sep 22. PMID 19772683
- [Background] Julvez J, Fortuny J, Mendez M, Torrent M, Ribas-Fito N, Sunyer J. Maternal use of folic acid supplements during pregnancy and four-year-old neurodevelopment in a population-based birth cohort. Paediatr Perinat Epidemiol. 2009 May;23(3):199-206. doi: 10.1111/j.1365-3016.2009.01032.x. Epub 2009 Mar 11. PMID 19775381
- [Background] Beard CM, Panser LA, Katusic SK. Is excess folic acid supplementation a risk factor for autism? Med Hypotheses. 2011 Jul;77(1):15-7. doi: 10.1016/j.mehy.2011.03.013. Epub 2011 Mar 31. PMID 21454018
- [Background] King CR. A novel embryological theory of autism causation involving endogenous biochemicals capable of initiating cellular gene transcription: a possible link between twelve autism risk factors and the autism 'epidemic'. Med Hypotheses. 2011 May;76(5):653-60. doi: 10.1016/j.mehy.2011.01.024. Epub 2011 Mar 8. PMID 21388746
- [Background] Salbaum JM, Kappen C. Genetic and epigenomic footprints of folate. Prog Mol Biol Transl Sci. 2012;108:129-58. doi: 10.1016/B978-0-12-398397-8.00006-X. PMID 22656376
- [Background] Fenech M. Folate (vitamin B9) and vitamin B12 and their function in the maintenance of nuclear and mitochondrial genome integrity. Mutat Res. 2012 May 1;733(1-2):21-33. doi: 10.1016/j.mrfmmm.2011.11.003. Epub 2011 Nov 7. PMID 22093367
- [Background] LaSalle JM. A genomic point-of-view on environmental factors influencing the human brain methylome. Epigenetics. 2011 Jul;6(7):862-9. doi: 10.4161/epi.6.7.16353. Epub 2011 Jul 1. PMID 21617367
- [Background] Chang CM, Yu CC, Lu HT, Chou YF, Huang RF. Folate deprivation promotes mitochondrial oxidative decay: DNA large deletions, cytochrome c oxidase dysfunction, membrane depolarization and superoxide overproduction in rat liver. Br J Nutr. 2007 May;97(5):855-63. doi: 10.1017/S0007114507666410. PMID 17381984
- [Background] Blaise SA, Alberto JM, Audonnet-Blaise S, Gueant JL, Daval JL. Influence of preconditioning-like hypoxia on the liver of developing methyl-deficient rats. Am J Physiol Endocrinol Metab. 2007 Dec;293(6):E1492-502. doi: 10.1152/ajpendo.00255.2007. Epub 2007 Aug 28. PMID 17726145
- [Background] Ferguson SA, Berry KJ, Hansen DK, Wall KS, White G, Antony AC. Behavioral effects of prenatal folate deficiency in mice. Birth Defects Res A Clin Mol Teratol. 2005 Apr;73(4):249-52. doi: 10.1002/bdra.20111. PMID 15744731
- [Background] Kerek R, Geoffroy A, Bison A, Martin N, Akchiche N, Pourie G, Helle D, Gueant JL, Bossenmeyer-Pourie C, Daval JL. Early methyl donor deficiency may induce persistent brain defects by reducing Stat3 signaling targeted by miR-124. Cell Death Dis. 2013 Aug 8;4(8):e755. doi: 10.1038/cddis.2013.278. PMID 23928694
- [Background] Moretti P, Sahoo T, Hyland K, Bottiglieri T, Peters S, del Gaudio D, Roa B, Curry S, Zhu H, Finnell RH, Neul JL, Ramaekers VT, Blau N, Bacino CA, Miller G, Scaglia F. Cerebral folate deficiency with developmental delay, autism, and response to folinic acid. Neurology. 2005 Mar 22;64(6):1088-90. doi: 10.1212/01.WNL.0000154641.08211.B7. PMID 15781839
- [Background] Amir RE, Van den Veyver IB, Wan M, Tran CQ, Francke U, Zoghbi HY. Rett syndrome is caused by mutations in X-linked MECP2, encoding methyl-CpG-binding protein 2. Nat Genet. 1999 Oct;23(2):185-8. doi: 10.1038/13810. PMID 10508514
- [Background] Neul JL. The relationship of Rett syndrome and MECP2 disorders to autism. Dialogues Clin Neurosci. 2012 Sep;14(3):253-62. doi: 10.31887/DCNS.2012.14.3/jneul. PMID 23226951
- [Background] Padmanabhan N, Jia D, Geary-Joo C, Wu X, Ferguson-Smith AC, Fung E, Bieda MC, Snyder FF, Gravel RA, Cross JC, Watson ED. Mutation in folate metabolism causes epigenetic instability and transgenerational effects on development. Cell. 2013 Sep 26;155(1):81-93. doi: 10.1016/j.cell.2013.09.002. PMID 24074862
- [Background] James SJ, Melnyk S, Jernigan S, Pavliv O, Trusty T, Lehman S, Seidel L, Gaylor DW, Cleves MA. A functional polymorphism in the reduced folate carrier gene and DNA hypomethylation in mothers of children with autism. Am J Med Genet B Neuropsychiatr Genet. 2010 Sep;153B(6):1209-20. doi: 10.1002/ajmg.b.31094. PMID 20468076
- [Background] Whitrow MJ, Moore VM, Rumbold AR, Davies MJ. Effect of supplemental folic acid in pregnancy on childhood asthma: a prospective birth cohort study. Am J Epidemiol. 2009 Dec 15;170(12):1486-93. doi: 10.1093/aje/kwp315. Epub 2009 Oct 30. PMID 19880541
- [Background] Crider KS, Cordero AM, Qi YP, Mulinare J, Dowling NF, Berry RJ. Prenatal folic acid and risk of asthma in children: a systematic review and meta-analysis. Am J Clin Nutr. 2013 Nov;98(5):1272-81. doi: 10.3945/ajcn.113.065623. Epub 2013 Sep 4. PMID 24004895
- [Background] Martinussen MP, Risnes KR, Jacobsen GW, Bracken MB. Folic acid supplementation in early pregnancy and asthma in children aged 6 years. Am J Obstet Gynecol. 2012 Jan;206(1):72.e1-7. doi: 10.1016/j.ajog.2011.07.033. Epub 2011 Jul 29. PMID 21982024
- [Background] Toriello HV; Policy and Practice Guideline Committee of the American College of Medical Genetics. Policy statement on folic acid and neural tube defects. Genet Med. 2011 Jun;13(6):593-6. doi: 10.1097/GIM.0b013e31821d4188. PMID 21552133
- [Background] Keating E, Goncalves P, Campos I, Costa F, Martel F. Folic acid uptake by the human syncytiotrophoblast: interference by pharmacotherapy, drugs of abuse and pathological conditions. Reprod Toxicol. 2009 Dec;28(4):511-20. doi: 10.1016/j.reprotox.2009.07.001. Epub 2009 Jul 16. PMID 19616087
- [Background] Cooney CA, Dave AA, Wolff GL. Maternal methyl supplements in mice affect epigenetic variation and DNA methylation of offspring. J Nutr. 2002 Aug;132(8 Suppl):2393S-2400S. doi: 10.1093/jn/132.8.2393S. PMID 12163699
- [Background] Waterland RA, Travisano M, Tahiliani KG, Rached MT, Mirza S. Methyl donor supplementation prevents transgenerational amplification of obesity. Int J Obes (Lond). 2008 Sep;32(9):1373-9. doi: 10.1038/ijo.2008.100. Epub 2008 Jul 15. PMID 18626486
- [Background] Wolff GL, Kodell RL, Moore SR, Cooney CA. Maternal epigenetics and methyl supplements affect agouti gene expression in Avy/a mice. FASEB J. 1998 Aug;12(11):949-57. PMID 9707167
- [Background] Mann JR, McDermott S, Bao H, Hardin J, Gregg A. Pre-eclampsia, birth weight, and autism spectrum disorders. J Autism Dev Disord. 2010 May;40(5):548-54. doi: 10.1007/s10803-009-0903-4. PMID 19936906
- [Background] Johnson S, Wolke D. Behavioural outcomes and psychopathology during adolescence. Early Hum Dev. 2013 Apr;89(4):199-207. doi: 10.1016/j.earlhumdev.2013.01.014. Epub 2013 Feb 27. PMID 23455605
- [Background] Movsas TZ, Paneth N. The effect of gestational age on symptom severity in children with autism spectrum disorder. J Autism Dev Disord. 2012 Nov;42(11):2431-9. doi: 10.1007/s10803-012-1501-4. PMID 22422339
- [Background] Asztalos EV, Murphy KE, Willan AR, Matthews SG, Ohlsson A, Saigal S, Armson BA, Kelly EN, Delisle MF, Gafni A, Lee SK, Sananes R, Rovet J, Guselle P, Amankwah K, Saleem M, Sanchez J; MACS-5 Collaborative Group. Multiple courses of antenatal corticosteroids for preterm birth study: outcomes in children at 5 years of age (MACS-5). JAMA Pediatr. 2013 Dec;167(12):1102-10. doi: 10.1001/jamapediatrics.2013.2764. PMID 24126948
- [Background] Constantino JN, Davis SA, Todd RD, Schindler MK, Gross MM, Brophy SL, Metzger LM, Shoushtari CS, Splinter R, Reich W. Validation of a brief quantitative measure of autistic traits: comparison of the social responsiveness scale with the autism diagnostic interview-revised. J Autism Dev Disord. 2003 Aug;33(4):427-33. doi: 10.1023/a:1025014929212. PMID 12959421
- [Background] Gioia GA. Isquith PK GP, Kenworthy L. Behavior Rating Inventory of Executive Function (BRIEF). Odessa, Fl: Psychological Assessment Resources, 2000.
- [Background] Achenbach TM, Dumenci, L., & Rescorla, L. A. Ten-Year Comparisons of Problems and Competencies for National Samples of Youth: Self, Parent, and Teacher Reports. Journal of Emotional and Behavioral Disorders 2002;10:194-203.
- [Background] Charman T, Baird G, Simonoff E, Loucas T, Chandler S, Meldrum D, Pickles A. Efficacy of three screening instruments in the identification of autistic-spectrum disorders. Br J Psychiatry. 2007 Dec;191:554-9. doi: 10.1192/bjp.bp.107.040196. PMID 18055961
- [Background] Bolte S, Dickhut H, Poustka F. Patterns of parent-reported problems indicative in autism. Psychopathology. 1999 Mar-Apr;32(2):93-7. doi: 10.1159/000029072. PMID 10026453
- [Background] Duarte CS, Bordin IA, de Oliveira A, Bird H. The CBCL and the identification of children with autism and related conditions in Brazil: pilot findings. J Autism Dev Disord. 2003 Dec;33(6):703-7. doi: 10.1023/b:jadd.0000006005.31818.1c. PMID 14714937
- [Background] Constantino JN, & Gruber, C. P. Social Responsiveness Scale (SRS): Manual. Los Angeles: Western Psychological Services, 2005.
- [Background] Wilkinson LA. A best practice guide to assessment and intervention for autism and Asperger syndrome in schools. London: Jessica Kingsley Publishers, 2010.
- [Background] Bolte S, Poustka F, Constantino JN. Assessing autistic traits: cross-cultural validation of the social responsiveness scale (SRS). Autism Res. 2008 Dec;1(6):354-63. doi: 10.1002/aur.49. PMID 19360690
- [Background] Fombonne E, Marcin C, Bruno R, Tinoco CM, Marquez CD. Screening for autism in Mexico. Autism Res. 2012 Jun;5(3):180-9. doi: 10.1002/aur.1235. Epub 2012 May 11. PMID 22581514
- [Background] Hsiao MN, Tseng WL, Huang HY, Gau SS. Effects of autistic traits on social and school adjustment in children and adolescents: the moderating roles of age and gender. Res Dev Disabil. 2013 Jan;34(1):254-65. doi: 10.1016/j.ridd.2012.08.001. Epub 2012 Sep 7. PMID 22960068
- [Background] Kamio Y, Moriwaki A, Inada N. Utility of teacher-report assessments of autistic severity in Japanese school children. Autism Res Treat. 2013;2013:373240. doi: 10.1155/2013/373240. Epub 2013 Dec 11. PMID 24392224
- [Background] Wigham S, McConachie H, Tandos J, Le Couteur AS; Gateshead Millennium Study core team. The reliability and validity of the Social Responsiveness Scale in a UK general child population. Res Dev Disabil. 2012 May-Jun;33(3):944-50. doi: 10.1016/j.ridd.2011.12.017. Epub 2012 Jan 25. PMID 22277583
- [Background] Constantino JNGC. Social Responsiveness Scale, Second Edition. Los Angeles: Western Psychological Services, 2012.
- [Background] Anderson P. Assessment and development of executive function (EF) during childhood. Child Neuropsychol. 2002 Jun;8(2):71-82. doi: 10.1076/chin.8.2.71.8724. PMID 12638061
- [Background] Gioia GA EK, & Isquith, PK. . Behavior Rating Inventory of Executive Function, Preschool Version. Lutz, Fl: Psychological Assessment Resources, Inc., 2003.
- [Background] Braun JM, Kalkbrenner AE, Calafat AM, Yolton K, Ye X, Dietrich KN, Lanphear BP. Impact of early-life bisphenol A exposure on behavior and executive function in children. Pediatrics. 2011 Nov;128(5):873-82. doi: 10.1542/peds.2011-1335. Epub 2011 Oct 24. PMID 22025598
- [Background] Duku E, Vaillancourt T. Validation of the BRIEF-P in a sample of Canadian preschool children. Child Neuropsychol. 2014;20(3):358-71. doi: 10.1080/09297049.2013.796919. Epub 2013 May 31. PMID 23721091
- [Background] Egeland J, Fallmyr O. Confirmatory Factor Analysis of the Behavior Rating Inventory of Executive Function (BRIEF): support for a distinction between emotional and behavioral regulation. Child Neuropsychol. 2010;16(4):326-37. doi: 10.1080/09297041003601462. Epub 2010 Mar 5. PMID 20209415
- [Background] Gioia GA, Isquith PK, Retzlaff PD, Espy KA. Confirmatory factor analysis of the Behavior Rating Inventory of Executive Function (BRIEF) in a clinical sample. Child Neuropsychol. 2002 Dec;8(4):249-57. doi: 10.1076/chin.8.4.249.13513. PMID 12759822
- [Background] Achenbach TM, & Rescorla, L.A. Manual for the ASEBA Preschool forms and Profiles. Burlington, VT: University of Vermont Department of Psychiatry, 2000.
- [Background] Achenbach T. Manual for the Child Behavior Checklist/2-1 and 1992 Profile. Burlington (VT): University of Vermont Department of Psychiatry, 1992.
- [Background] Achenbach TM, & Rescorla, L. A. Manual for the ASEBA School-Age Forms & Profiles. Burlington, VT: University of Vermont, Research Center for Children, Youth, & Families, 2001.
- [Background] Cai X, Kaiser AP, Hancock TB. Parent and teacher agreement on child behavior checklist items in a sample of preschoolers from low-income and predominantly African American families. J Clin Child Adolesc Psychol. 2004 Jun;33(2):303-12. doi: 10.1207/s15374424jccp3302_12. PMID 15136195
- [Background] Pandolfi V, Magyar CI, Dill CA. Confirmatory factor analysis of the child behavior checklist 1.5-5 in a sample of children with autism spectrum disorders. J Autism Dev Disord. 2009 Jul;39(7):986-95. doi: 10.1007/s10803-009-0716-5. Epub 2009 Mar 5. PMID 19263208
- [Background] Suglia SF, Duarte CS, Chambers EC, Boynton-Jarrett R. Social and behavioral risk factors for obesity in early childhood. J Dev Behav Pediatr. 2013 Oct;34(8):549-56. doi: 10.1097/DBP.0b013e3182a509c0. PMID 24131877
- [Background] Tan TX, Dedrick RF, Marfo K. Factor structure and clinical implications of child behavior checklist/1.5-5 ratings in a sample of girls adopted from China. J Pediatr Psychol. 2007 Aug;32(7):807-18. doi: 10.1093/jpepsy/jsm025. Epub 2007 Apr 19. PMID 17449465
- [Background] Austin PC, Lee DS, Fine JP. Introduction to the Analysis of Survival Data in the Presence of Competing Risks. Circulation. 2016 Feb 9;133(6):601-9. doi: 10.1161/CIRCULATIONAHA.115.017719. PMID 26858290
- [Background] AP Association. Diagnostic and statistical manual of mental disorders (5th Ed.). Washington, DC.: American Psychiatric Publishing, 2013.
- [Background] Andrews, D. Children With School Problems: A Physician's Manual: The Canadian Paediatric Society, 2012.